CLINICAL TRIAL: NCT01090739
Title: An Investigation of the Treatment of Fecal Incontinence Using the TOPAS Sling System For Women (TRANSFORM)
Brief Title: Clinical Study to Investigate the Effectiveness of the TOPAS System to Treat Fecal Incontinence
Acronym: TRANSFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASTORA Women's Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WC0807
Record Dates: First submitted 2010-03-19; First posted 2010-03-22 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Accidental bowel leakage; Failure conservative therapy; Women; Class III medical device; Surgical mesh
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TOPAS (Experimental): TOPAS Treatment for Fecal Incontinence
  Interventions: Device: TOPAS Treatment for Fecal Incontinence

INTERVENTIONS:
Device: TOPAS Treatment for Fecal Incontinence — The TOPAS Treatment for Fecal Incontinence is implanted using a minimally invasive trans-obturator approach; two needle passers deliver the sling assembly. Two small posterior incisions facilitate the post-anal placement of the mesh.

SUMMARY:
The purpose of this study is to demonstrate that the TOPAS System effectively treats fecal incontinence in women as measured by a 50% reduction in the number of FI episodes in a 14 day bowel diary at 12 months.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm, open-label, two- stage, adaptive study conducted to obtain data to demonstrate the safety and effectiveness of the TOPAS system for the treatment of FI in women who have failed conservative therapy. It was approved by the FDA for up to 152 implanted subjects at up to 15 investigational sites in the US. Eight study centers are led by a Colorectal Surgeon and seven centers are led by an Urogynecologist.

This study is being conducted in compliance with Title 21 CFR Parts 11, 50, 54, 56, and 812; the principles of GCP as set forth in the World Medical Association Declaration of Helsinki (2008); and the ISO standard 14155:2011 (Clinical investigation of medical devices for human subjects - Good clinical practice).

ELIGIBILITY:
Inclusion Criteria:

Subject is/has:

1. An adult (>/= 18 years) female.
2. FI symptoms for a minimum of 6 months.
3. Failed two modalities of conservative therapies such as Dietary Modification, Pharmacologic Intervention, or Pelvic Floor Muscle Training.
4. <50 years old OR if >/= 50 years old, has had a negative cancer screening examination of the colon according screening guidelines (colonoscopy or barium enema + flexible sigmoidoscopy) within the past 3 years prior to informed consent date. (Note: if not done, the investigating physician must provide written justification for not having this exam and must be following the American Cancer Society Guidelines).
5. FI episodes ≥ 4 in 14 day period.

Exclusion Criteria:

Subject is/has

1. Unable or unwilling to sign Informed Consent Form or comply with study requirements.
2. Currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study as determined by AMS.
3. Allergic to polypropylene.
4. Pregnant or planning a future pregnancy.
5. Less than 12 months (365 days) postpartum.
6. Pelvic prolapse >/=1 cm beyond the hymen (Stage III & IV)
7. Had stress urinary incontinence (SUI) or anterior repair within 3 months (90 days) prior to TOPAS Sling System implantation.
8. Had a hysterectomy, Sphincteroplasty, or Posterior surgery within 6 months (180 days) prior to TOPAS Sling System implantation.
9. Had rectal surgery (such as rectopexy) within 12 months (365 days) of TOPAS Sling System implantation.
10. Planning pelvic surgery within 12 months (365 days) post implant
11. Current Grade III or IV hemorrhoids.
12. Neurological or psychological condition as cause of FI such as MS, dementia, brain tumor.
13. Diagnosed Inflammatory Bowel Disease (for example, ulcerative colitis or Crohn's disease).
14. Chronic, watery diarrhea, unmanageable by drugs or diet, as primary cause of fecal incontinence.
15. Severe chronic constipation, including obstructive defecatory disorder.
16. External full thickness rectal prolapse.
17. A history of laxative abuse within the past 5 years.
18. Had previous rectal resection.
19. Active pelvic infection, perianal or recto-vaginal fistula.
20. Congenital anorectal malformations or chronic 4th degree lacerations and cloacae.
21. History of therapeutic radiation for cancers of the pelvis.
22. Currently implanted with a sacral nerve stimulator.
23. Contraindicated for surgery or having any condition that would compromise wound healing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2010-04; Primary Completion 2013-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Mellgren, MD, PhD, Study Chair — University of Illinois at Chicago; Dee Fenner, MD, Study Chair — University of Michigan
Locations (14):
- United States (14):
  - University of California SF - Mt Zion Medical Center, San Francisco, California
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Foundation - Florida, Weston, Florida
  - Raybon OB-GYN, Toccoa, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Atlantic Health System, Morristown, New Jersey
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation - Ohio, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - St. Luke's Hospital, Allentown, Pennsylvania
  - Womens Hospital of Texas, Houston, Texas
  - Sacred Heart Medical Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Each site was provided with their individual participant data

REFERENCES:
- [Result] Mellgren A, Zutshi M, Lucente VR, Culligan P, Fenner DE; TOPAS Study Group. A posterior anal sling for fecal incontinence: results of a 152-patient prospective multicenter study. Am J Obstet Gynecol. 2016 Mar;214(3):349.e1-8. doi: 10.1016/j.ajog.2015.10.013. Epub 2015 Oct 19. PMID 26493933
- See also: Primary (1 Year) Results Manuscript — http://dx.doi.org/10.1016/j.ajog.2015.10.013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred from July 2010 - December 2012.
Pre-assignment Details: Following enrollment (i.e., signing informed consent form), subjects underwent two screening visits to evaluate and confirm eligibility for the TOPAS implant procedures.
Period: Enrollment
Arm/Group | TOPAS
Started | 207 (Subject enrollment = signed informed consent form)
Completed | 152
Not Completed | 55
Not completed — Withdrawal by Subject | 24
Not completed — Protocol Violation | 14
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 5
Not completed — Sponsor termination of site | 4
Not completed — Study implant limit reached | 2
Not completed — Adverse Event | 1
Period: 12 Month Follow-up
Arm/Group | TOPAS
Started | 152
Completed | 147
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Death | 1
Period: 24 Month Follow-up
Arm/Group | TOPAS
Started | 147
Completed | 138
Not Completed | 9
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Period: 36 Month Follow-up
Arm/Group | TOPAS
Started | 138
Completed | 115
Not Completed | 23
Not completed — Withdrawal by Subject | 6
Not completed — Visit still pending | 17

BASELINE CHARACTERISTICS:
Population: All subjects who met the study inclusion/exclusion criteria and were implanted with the TOPAS device.
Arm/Group | TOPAS
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.7)
Sex/Gender, Customized [Number; unit: participants]
  Women | 152
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 137
  Black or African American | 10
  Asian | 1
  Hispanic/Latina | 3
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 152
Obstetric History - Gravidity [Mean (Standard Deviation); unit: number] — Number of times subjects have been pregnant
  number | 3.0 (1.8)
Obstetric History - Parity [Mean (Standard Deviation); unit: number] — Parity is defined as the number of pregnancies carried to gestation
  number | 2.6 (1.4)
Obstetric History - # of Vaginal Deliveries [Mean (Standard Deviation); unit: number] — The number of times a women delivered vaginally
  number | 2.4 (1.5)
Obstetric History - # of Caesarean deliveries [Mean (Standard Deviation); unit: number] — women delivering via a caesarean procedure
  number | 0.1 (0.5)
Menopausal Status [Number; unit: participants]
  Pre-menopausal | 20
  Peri-menopausal | 6
  Post-menopausal | 126
Concomitant Use [Number; unit: participants]
  # Smoked within past 6 months | 8
  # Caffeine use on a regular basis | 102
  # Rgular laxative use within past 5 years | 18
Duration of Fecal Incontinence [Mean (Standard Deviation); unit: months] | 110.0 (113.5)
Etiology of Fecal Incontinence [Number; unit: participants] — Subjects can have multiple etiologies so total does not equal 152 (number of subjects)
  participants
    Anorectal trauma | 6
    Obstetric trauma | 87
    Idiopathic/unknown | 62
    Other | 4
Rectal soft tissue scarring [Number; unit: participants]
  Present | 26
  Absent | 126
Baseline Medical History [Number; unit: participants] — Subjects can have multiple medical history items so the total does not equal 152 (number of subjects).
  participants
    Previous hysterectomy / oophorectomy | 74
    Previous prolapse / UI repair | 70
    Gastrointestional reflux disease | 65
    Hypertension | 60
    Depressive disorder | 56
    Systemic pain | 55
    Hyperlipidemia | 53
    Pelvic area pain | 52
    Diverticulitis | 41
    Urinary incontinence | 39
    Hypothroid | 38
    Previous cholecystectomy | 38
    Hemorrhoids | 36
    Irritable bowel syndrome | 31
    Previous anal sphincter repair | 31
    Headaches | 29
    Vaginal atrophy | 23
    Diabetes | 19
    Vaginal prolapse | 8
    Rectal prolapse | 6
    Gallstones | 2
Baseline Fecal Incontinence Medication [Number; unit: participants] — Subjects taking medications does not equal 152 (number of subjects).
  participants
    Opioid-receptor agents | 30
    Bulking agents | 22
    Osmotic laxatives | 8
    Anti-cholinergic agents | 6
    Other meds | 5
    Bile acid sequestrants | 3
Failed Fecal Incontinence Conservative Therapy [Number; unit: participants] — Subjects had to fail at least two conservative therapies for their FI prior to entry into the study.
  participants
    Diet modification and medication | 22
    Diet modification and pelvic floor muscle training | 49
    Medication and pelvic floor muscle training | 20
    Diet, medication and pelvic floor training | 61
Hemorrhoids [Number; unit: participants]
  Present | 34
  Absent | 118
Anal Resting Tone [Number; unit: participants]
  Present | 141
  Absent | 11
Anorectal Manometry - Pressures [Mean (Standard Deviation); unit: mmHg]
  Mean Maximum Resting Pressure | 31.5 (21.9)
  Mean Maximum Squeeze Pressure | 60.1 (42.6)
Anorectal Manometry - Volumes [Mean (Standard Deviation); unit: cc]
  First sensation volume | 43.1 (30.9)
  Maximum tolerated volume | 124.8 (61.9)
External Anal Sphincter Defects [Number; unit: participants]
  Present | 79
  Absent | 73
Internal Anal Sphincter Defects [Number; unit: participants]
  Present | 42
  Absent | 110
External Anal Sphincter Defect Extent [Mean (Standard Deviation); unit: degrees] | 95.3 (45.0)
Internal Anal Sphincter Defect Extent [Mean (Standard Deviation); unit: degrees] | 110.0 (53.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: The primary endpoint for efficacy is the 14 day bowel diary documenting liquid or solid fecal incontinence episodes. A 50% reduction in the number of FI episodes is considered a treatment responder.
Time Frame: 12 Months
Population: All subjects implanted
Measure: Number (95% Confidence Interval); unit: percentage of treatment responders
Arm/Group | TOPAS
Number analyzed (Participants) | 152
percentage of treatment responders | 69.1 [61.1 to 76.3]

2. Secondary Outcome: Change in Fecal Incontinence Episodes
Description: Number of fecal incontinence episodes in a 14 day period
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Median (Full Range); unit: fecal incontinent episodes/14 days
Arm/Group | TOPAS
Number analyzed (Participants) | 152
fecal incontinent episodes/14 days
  Baseline | 18 [4 to 81]
  3 Months | 5 [0 to 94]
  6 Months | 5 [0 to 67]
  12 Months | 5 [0 to 80]
  24 Months | 5 [0 to 73]
  36 Months | 5 [0 to 52]

3. Secondary Outcome: Change in Fecal Incontinence Days
Description: Number of fecal incontinence days in a 14 day period
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Median (Full Range); unit: fecal incontinent days/14 days
Arm/Group | TOPAS
Number analyzed (Participants) | 152
fecal incontinent days/14 days
  Baseline | 10 [3 to 14]
  3 Months | 4 [0 to 14]
  6 Months | 4 [0 to 14]
  12 Months | 4 [0 to 14]
  24 Months | 4 [0 to 14]
  36 Months | 4 [0 to 14]

4. Secondary Outcome: Change in Urge Fecal Incontinence Episodes
Description: Number of urge fecal incontinence episodes in a 14 day period
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Median (Full Range); unit: urge fecal incontinent episodes/14 days
Arm/Group | TOPAS
Number analyzed (Participants) | 152
urge fecal incontinent episodes/14 days
  Baseline | 4 [0 to 52]
  3 Months | 0 [0 to 16]
  6 Months | 0 [0 to 18]
  12 Months | 0 [0 to 29]
  24 Months | 0 [0 to 39]
  36 Months | 0 [0 to 34]

5. Secondary Outcome: Change in Wexner Symptom Severity Score
Description: Wexner Symptom Severity Score for fecal incontinence (also known as the Cleveland Clinic Incontinence Score) as described by Jorge and Wexner, 1993 (Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97). Measured on a 0-20 scale with lower scores equal to less fecal incontinence.
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 152
units on a scale
  Baseline | 13.9 (2.7)
  3 Months | 9.4 (4.3)
  6 Months | 9.8 (4.4)
  12 Months | 9.6 (3.9)
  24 Months | 9.5 (4.2)
  36 Months | 9.4 (4.3)

6. Secondary Outcome: Change in Fecal Incontinence Quality of Life Score
Description: Fecal Incontinence Quality of Life Score as described by Rockwood et al., 2000 (Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7). Four domains of lifestyle, coping, depression, and embarrassment. Measured on a 0-4 scale with higher scores equal to better quality of life.
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 152
units on a scale
  Lifestyle - Baseline | 2.6 (0.8)
  Lifestyle - 3 Months | 3.3 (0.7)
  Lifestyle - 6 Months | 3.3 (0.7)
  Lifestyle - 12 Months | 3.4 (0.7)
  Lifestyle - 24 Months | 3.4 (0.7)
  Lifestyle - 36 Months | 3.4 (0.7)
  Coping - Baseline | 1.7 (0.6)
  Coping - 3 Months | 2.6 (0.8)
  Coping - 6 Months | 2.6 (0.9)
  Coping - 12 Months | 2.7 (0.9)
  Coping - 24 Months | 2.7 (0.9)
  Coping - 36 Months | 2.7 (0.9)
  Depression - Baseline | 2.4 (0.6)
  Depression - 3 Months | 3.0 (0.7)
  Depression - 6 Months | 3.1 (0.7)
  Depression - 12 Months | 3.1 (0.7)
  Depression - 24 Months | 3.1 (0.7)
  Depression - 36 Months | 3.2 (0.7)
  Embarrassment - Baseline | 1.6 (0.6)
  Embarrassment - 3 Months | 2.5 (0.9)
  Embarrassment - 6 Months | 2.6 (1.0)
  Embarrassment - 12 Months | 2.7 (0.9)
  Embarrassment - 24 Months | 2.7 (0.9)
  Embarrassment - 36 Months | 2.7 (0.9)

7. Secondary Outcome: Change in Pelvic Floor Distress Inventory (PFDI-20) Scores
Description: Short-form version of the Pelvic Floor Distress Inventory (PFDI-20) as described by Barber et al., 2005 (Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7. Am J Obstet Gynecol. 2005 Jul;193(1):103-13).
  The short-form version of the Pelvic Floor Distress Inventory has a total of 20 questions and 3 scales (Urinary Distress Inventory, Pelvic Organ Prolapse Distress Inventory, and Colorectal-Anal Distress Inventory). Total PFDI score measured on a 0-300 scale with higher scores equal to greater pelvic floor distress. As with the Total PFDI Score, higher subscale scores equal greater pelvic floor distress, on a 0-100 scale.
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 152
units on a scale
  Total PFDI Score - Baseline | 104.1 (47.4)
  Total PFDI Score - 3 Months | 69.7 (43.1)
  Total PFDI Score - 6 Months | 68.8 (45.9)
  Total PFDI Score - 12 Months | 66.7 (43.4)
  Total PFDI Score - 24 Months | 65.7 (43.9)
  Total PFDI Score - 36 Months | 70.3 (51.2)
  Colorectal-Anal Subscale - Baseline | 54.8 (16.2)
  Colorectal-Anal Subscale - 3 Months | 33.3 (17.7)
  Colorectal-Anal Subscale - 6 Months | 33.0 (19.8)
  Colorectal-Anal Subscale - 12 Months | 32.1 (19.2)
  Colorectal-Anal Subscale - 24 Months | 31.5 (19.7)
  Colorectal-Anal Subscale - 36 Months | 33.5 (21.0)
  Urinary Subscale - Baseline | 27.2 (25.1)
  Urinary Subscale - 3 Months | 21.4 (21.5)
  Urinary Subscale - 6 Months | 21.4 (22.7)
  Urinary Subscale - 12 Months | 21.5 (21.9)
  Urinary Subscale - 24 Months | 22.2 (22.1)
  Urinary Subscale - 36 Months | 22.6 (23.0)
  POP Subscale - Baseline | 21.9 (19.5)
  POP Subscale - 3 Months | 14.9 (15.6)
  POP Subscale - 6 Months | 14.2 (14.9)
  POP Subscale - 12 Months | 12.8 (13.9)
  POP Subscale - 24 Months | 12.1 (13.8)
  POP Subscale - 36 Months | 13.8 (16.9)

8. Secondary Outcome: Change in Pelvic Floor Impact Questionnaire (PFIQ-7) Scores
Description: Short-form version of the Pelvic Floor Impact Questionnaire (PFIQ-7) as described by Barber et al., 2005 (Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7. Am J Obstet Gynecol. 2005 Jul;193(1):103-13).
  The short-form version of the Pelvic Floor Impact Questionnaire has a total of 7 questions and 3 scales (Urinary Impact, Pelvic Organ Prolapse Impact, and Colorectal-Anal Impact). Total PFIQ score measured on a 0-300 scale with higher scores equal to greater pelvic floor impact. Subscales scored on 0-100 scale and the higher the score the greater pelvic floor impact, exactly like the Total PFIQ score.
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 152
units on a scale
  Total PDFI Score - Baseline | 79.6 (52.3)
  Total PDFI Score - 3 Months | 41.0 (43.5)
  Total PDFI Score - 6 Months | 39.6 (48.4)
  Total PDFI Score - 12 Months | 37.9 (43.5)
  Total PDFI Score - 24 Months | 35.2 (45.5)
  Total PDFI Score - 36 Months | 38.5 (48.5)
  Colorectal-Anal Subscale - Baseline | 51.7 (25.5)
  Colorectal-Anal Subscale - 3 Months | 23.1 (22.7)
  Colorectal-Anal Subscale - 6 Months | 23.3 (24.1)
  Colorectal-Anal Subscale - 12 Months | 21.7 (22.6)
  Colorectal-Anal Subscale - 24 Months | 20.4 (22.9)
  Colorectal-Anal Subscale - 36 Months | 20.9 (22.1)
  Urinary Subscale - Baseline | 18.5 (23.6)
  Urinary Subscale - 3 Months | 12.7 (19.8)
  Urinary Subscale - 6 Months | 10.8 (18.3)
  Urinary Subscale - 12 Months | 11.3 (18.1)
  Urinary Subscale - 24 Months | 10.4 (17.7)
  Urinary Subscale - 36 Months | 11.8 (19.6)
  POP Subscale - Baseline | 9.8 (19.5)
  POP Subscale - 3 Months | 5.2 (11.8)
  POP Subscale - 6 Months | 5.8 (16.3)
  POP Subscale - 12 Months | 4.8 (12.7)
  POP Subscale - 24 Months | 4.5 (13.9)
  POP Subscale - 36 Months | 5.8 (14.5)

9. Secondary Outcome: Change in Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12)
Description: Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) as described by Rogers RG, Coates KW, Kammerer-Doak D, Khalsa S, Qualls C. A short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J Pelvic Floor Dysfunct. 2003 Aug;14(3):164-8; discussion 168. Measured on a 0-48 scale with higher scores equal to better sexual function.
Time Frame: 36 Month Follow-up Visit
Population: All subjects implanted
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 152
units on a scale
  Baseline | 32.2 (6.7)
  3 Months | 35.1 (6.1)
  6 Months | 35.0 (6.9)
  12 Months | 34.6 (7.1)
  24 Months | 33.9 (7.9)
  36 Months | 35.1 (7.8)

10. Secondary Outcome: Change in Numeric Pelvic Pain Scale (NPPS)
Description: Numeric Pelvic Pain Scale (NPPS) adapted from McCafferty M, Pasero C. Pain: Clinical Manual. 2nd ed. Philadelphia: Mosby Inc.; 1999. Chapter 3, Assessment Tools; p. 58-75. The NPPS is scored on a 0-10 scale with higher scores indicating more severe pain. Since the NPPS was introduced later in the study, earlier implanted subjects did not have the baseline NPPS score and a change from baseline could not be calculated.
Time Frame: 12 Month Follow-up Visit
Population: All subjects implanted at the time the NPPS was implemented in the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 103
units on a scale
  Baseline | 0.8 (1.7)
  Procedure | 3.2 (2.5)
  Acute Follow-up | 1.0 (1.9)
  3 Months | 0.4 (1.1)
  6 Months | 0.7 (1.8)
  12 Months | 0.6 (1.6)

11. Other Pre Specified Outcome: Change in the Haff Surgical Satisfaction Questionnaire (SSQ-8)
Description: The SSQ-8 is an 8 item questionnaire to assess subject surgical satisfaction as described by Murphy M, Sternschuss G, Haff R, van Raalte H, Saltz S, Lucente V. Quality of life and surgical satisfaction after vaginal reconstructive vs. obliterative surgery for the treatment of advanced pelvic organ prolapse. Am J Obstet Gynecol. 2008 May;198(5):573.e1-7. The SSQ-8 was collected as an optional one-time assessment from implanted subjects between the 3 and 36 month visits. Scale is scored on 0-100 with higher scores are better
Time Frame: 36 Month Follow-up Visit
Population: All implanted subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOPAS
Number analyzed (Participants) | 86
units on a scale | 79.4 (22.1)

12. Other Pre Specified Outcome: Change in Health Resource Usage: # Pads Per Day Subject Took for FI
Description: Change in health resource usage using sponsor-created questionnaire: # days in hospital due to FI
Time Frame: 36 Month Follow-up Visit
Population: All implanted subjects
Measure: Mean (Standard Deviation); unit: pads per day
Arm/Group | TOPAS
Number analyzed (Participants) | 152
pads per day
  # pads per day subject took for FI - Baseline | 2.4 (2.1)
  # per day subject took for FI - 12 Months | 1.4 (1.8)
  # pads per day subject took for FI - 24 Months | 1.1 (1.5)
  # pads per day subject took for FI - 36 Months | 1.2 (1.6)

13. Other Pre Specified Outcome: Change in Health Resource Usage: # Days in Hospital, Took Off Work, or Others Took Off Work Due to FI
Description: Change in health resource usage using sponsor-created questionnaire
Time Frame: 36 Month Follow-up Visit
Population: All implanted subjects
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TOPAS
Number analyzed (Participants) | 152
days
  # days in hospital due to FI - Baseline | 0.1 (0.6)
  # days in hospital due to FI - 12 Months | 0.1 (0.5)
  # days in hospital due to FI - 24 Months | 0.0 (0.1)
  # days in hospital due to FI - 36 Months | 0.0 (0.0)
  # days took off work due to FI - Baseline | 6.4 (34.0)
  # days took off work due to FI - 12 Months | 1.3 (9.9)
  # days took off work due to FI - 24 Months | 4.5 (35.4)
  # days took off work due to FI - 36 Months | 0.9 (9.5)
  # days others took off work - Baseline | 0.2 (1.3)
  # days others took off work - 12 Months | 0.0 (0.0)
  # days others took off work - 24 Months | 0.0 (0.3)
  # days others took off work - 36 Months | 0.0 (0.0)

14. Other Pre Specified Outcome: Change in Health Resource Usage: # Physician Visits Due to FI
Description: Change in health resource usage using sponsor-created questionnaire
Time Frame: 36 Month Follow-up Visit
Population: All implanted subjects
Measure: Mean (Standard Deviation); unit: physician visits
Arm/Group | TOPAS
Number analyzed (Participants) | 152
physician visits
  # physician visits due to FI - Baseline | 5.0 (7.6)
  # physician visits due to FI - 12 Months | 0.4 (1.4)
  # physician visits due to FI - 24 Months | 0.5 (1.8)
  # physician visits due to FI - 36 Months | 0.3 (1.1)

ADVERSE EVENTS:
Time Frame: AEs collected for each subject from the time of enrollment (signing informed consent form) through duration of follow-up visits (up to 60 months). The mean follow-up period for all subjects was 40.2 months (509 subject years).
Description: An independent Adverse Event Adjudication Committee (three physicians: Colorectal, Gastroenterology, Urogynecology) reviewed all AEs and death data and assigned or verified correct assignment of codes, event seriousness, relatedness to the study device and/or procedure. All AEs listed here are device- and/or procedure-related only.
Arm/Group | TOPAS
Serious Adverse Events (participants affected / at risk) | 8/152
Other Adverse Events (participants affected / at risk) | 72/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOPAS (N=152)
Pain/discomfort - buttock (Musculoskeletal and connective tissue disorders) | 1 (1) — Exacerbation of sciatic pain
Worsening Pelvic Organ Prolapse (Reproductive system and breast disorders) | 1 (1) — Recurrent rectal prolapse
De novo pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) — Mild cystocele / enterocele / rectocele
Exacerbated post traumatic stress disorder (Psychiatric disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Worsening chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
De novo rectal prolapse (Reproductive system and breast disorders) | 1 (1) — Mucosal prolapse
Methicillin-resistant staphylococcus aureus infection (Infections and infestations) | 1 (1) — Hospital acquired - Left hand
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOPAS (N=152)
Pelvic area pain (Reproductive system and breast disorders) | 43 (50) — Pain/discomfort in the general pelvic region including the buttocks, groin, pelvis, upper leg, urogenitals and abdomen.
Infection (Infections and infestations) | 22 (25) — Includes incision site infection, abscess, UTIs, and fungal infections
Urinary problems (Renal and urinary disorders) | 8 (8) — Includes de novo and worsening urinary incontinence and retention
Pelvic organ prolapse (Reproductive system and breast disorders) | 9 (13) — Includes de novo and worsening vaginal and rectal prolapse
Bleeding (Injury, poisoning and procedural complications) | 1 (1)
Defecatory problems (Gastrointestinal disorders) | 4 (4) — includes worsening fecal incontinence and constipation
Other (Injury, poisoning and procedural complications) | 14 (14) — Includes Allergic Reaction / Hypersensitivity Reaction, Diarrhea, Headache, Deep Venous Thrombosis, COPD, Nausea, Post-Traumatic Stress Disorder, Rectal Discharge, Skin Irritation, and Wound Dehiscence

LIMITATIONS AND CAVEATS:
Study was a single arm trial with no control group. Study was done with a very specialized group of clinical investigators from two medical sub-specialties, Colorectal Surgeons and Urogynecologists. Study population was primarily Caucasian (90%).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the primary or the combined data article has been published, an Investigator may publish the study experience from his/her site. However, the Sponsor reserves the right to review the manuscript prior to submission in order to verify accuracy of the data.

All publications will be reviewed by the sponsor in order to assure that no confidential information is disclosed. Such confidential information is not allowed for publishing.